CLINICAL TRIAL: NCT01174706
Title: Impact of Information Prescriptions on Medication Adherence in ED Patients
Brief Title: Impact of Information Prescriptions on Medication Adherence in Emergency Department (ED) Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Library of Medicine (NLM) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: NA_00038209; 1RC1LM010424-01 (NIH)
Record Dates: First submitted 2010-08-03; First posted 2010-08-04 (Estimated); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Patient Compliance; Medication Adherence; Medication Non-Adherence
Keywords: infections; flu; abdominal pain; chest pain; cold; fever; different acute care conditions
MeSH Terms: conditions — Patient Compliance; Medication Adherence; Infections; Influenza, Human; Abdominal Pain; Chest Pain; Common Cold; Fever

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Usual care arm (Experimental): Patients randomized to this group will receive usual care. Usual care at the three study sites varies but will be defined as whatever information is usually given to patients regarding the prescription medication or over the counter medicine they were prescribed at emergency department discharge.
  Interventions: Behavioral: Information prescriptions
- Information prescription (Experimental): Patients randomized to this arm will receive written information from Medline Plus regarding the prescription or over the counter medicine they have been prescribed at ED discharge plus information on their health condition.
  Interventions: Behavioral: Information prescriptions
- Informationist (Experimental): Patients in this arm will receive the same information as patients in group 2 but will also be given contact information for a clinical informationist if they have further questions about their prescription medicine or over the counter medicine prescribed at ED discharge.
  Interventions: Behavioral: Information prescriptions
- practical assistance (Experimental): Subjects will be offered practical assistance with obtaining prescription such as location of most convenient pharmacy and hours of operation, programs that offer drugs more cheaply, fax prescription from ED to pharmacy
  Interventions: Behavioral: Information prescriptions

INTERVENTIONS:
Behavioral: Information prescriptions — One arm will receive usual care at discharge. The other three arms will receive practical assistance and/or an information prescription which will consist of written information from Medline Plus and access to a clinical informationist if subject has additional information needs.

SUMMARY:
The main objectives of this research are:

1. To identify factors that influence medication adherence rates in Emergency Department (ED) patients.
2. To measure the effects of alternative information prescriptions on medication adherence rates of ED patients.
3. To measure the effects of alternative information prescriptions (IRxs) on health and service utilization.

DETAILED DESCRIPTION:
People who are prescribed self-administered medications frequently take less than half the doses. Poor adherence to medication regimens is associated with worsening of disease, death and increased health care costs in the United States. The few studies conducted in the emergency department (ED) setting suggest that between 7 to 45 percent of patients do not fill their prescription; one study conducted in Canada reported that 45% of ED patients did not follow their prescribed regimen. One strategy that may improve medication adherence among ED patients is a better information exchange between the patient, provider and the health care system. This study will use a randomized controlled trial to test the effect that two alternative ways of delivering information prescriptions (IRxs) have on medication adherence and treatment outcomes of ED patients.

ED patients treated and released with a prescribed medication(s) from three hospitals serving different patient populations in the Baltimore metropolitan area over a 9 month period will be included in the study. Research assistants will consent eligible patients, interview them prior to ED discharge and randomize subjects to one of four study groups: (1) usual care (medication prescription and instructions provided at discharge); (2) practical assistance which consists of giving information to help subject obtain medicine (i.e. programs that offer drugs more cheaply, pharmacy hours of operation, etc)(3) an IRx that includes a MedlinePlus referral plus written information from MedlinePlus customized to the subject's health problem and prescribed medication; or (4) an IRx that consists of practical assistance and MedlinePlus referral plus customized written information from MedlinePlus plus access to information services provided by a medical librarian, herein referred to as a clinical informationist or informationist. Subjects will be contacted by telephone one week post ED visit and queried about medication use and patient outcomes (self-reported health, satisfaction with ED visit, and ED revisits or hospitalizations) and use of Internet to access health information. Medication instructions and ED discharge diagnosis data will be extracted from subjects' electronic medical record and use of informationist services documented. Medication adherence rates and patient outcomes will be compared among study groups. Self-reported use of MedlinePlus will also be compared to electronic data for all subjects. Self-reported medication and ED revisits/hospitalizations will be compared to pharmacy claims and utilization data for subjects covered by Medicaid.

ELIGIBILITY:
Inclusion Criteria: The study population will consist of adult patients who present to one of these three EDs during a 6 - 9 month period and are discharged with a medication regimen, either a prescription or over the counter (OTC) medication.

-

Exclusion Criteria: Patients will be excluded for the following reasons: (1) less than 18 years of age at time of ED visit; (2) non English or non Spanish speaking; (3) unable to understand consent or complete the baseline interview for cognitive, psychiatric or substance abuse reasons.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3940 (Actual)
Dates: Start 2010-11; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Medication adherence | one week after index ED visit
  Self-reported medication adherence.For subjects discharged with a prescription medication or an over the counter (OTC) medication with a specified dosage and frequency, medication adherence will be measured by the number of doses taken divided by the number of doses specified.

SECONDARY OUTCOMES:
Filling of prescription medicine | within one week of index ED visit
  This outcome will measure whether a patient filled the medication he was prescribed at ED discharge .

CONTACTS AND LOCATIONS:
Overall Officials: Melissa L McCarthy, ScD, Principal Investigator — Associate Professor; Nancy Roderer, MLS, Principal Investigator — Professor and Director of the Welch Medical Library
Locations (3):
- United States (3):
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Howard County General Hospital, Columbia, Maryland

REFERENCES:
- [Result] McCarthy ML, Ding R, Roderer NK, Steinwachs DM, Ortmann MJ, Pham JC, Bessman ES, Kelen GD, Atha W, Retezar R, Bessman SC, Zeger SL. Does providing prescription information or services improve medication adherence among patients discharged from the emergency department? A randomized controlled trial. Ann Emerg Med. 2013 Sep;62(3):212-23.e1. doi: 10.1016/j.annemergmed.2013.02.002. Epub 2013 Apr 3. PMID 23561463